CLINICAL TRIAL: NCT02793518
Title: Self-defining Memories and Future Projections in Bipolar Disorder Patients
Brief Title: Mental Time Travel and Identity in Bipolar Disorder Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Model: Parallel | Masking: None
Other Study IDs: PA12064
Record Dates: First submitted 2016-05-12; First posted 2016-06-08 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-05

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Psychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bipolar Disorder patients (Experimental)
  Interventions: Behavioral: psychological tests
- Healthy Controls (Experimental)
  Interventions: Behavioral: psychological tests

INTERVENTIONS:
Behavioral: psychological tests

SUMMARY:
Self-defining memories (SDMs) are memories that are still important today to understand who the investigators are and participate to the maintain of personal identity. SDMs are also linked to our capacity to project ourselves into the future. In bipolar disorder, life events play an important role in the course and outcome of the disease. the study is the first to investigate SDMs and self-defining future projections in a population of remitted patients with bipolar disorder.

DETAILED DESCRIPTION:
Study design: case / control study in inclusion prospective, single center. population:

* A group of 30 patients aged 18 to 60 years and followed in the psychiatry department of adult CHU Reims for bipolar disorder type I (DSM-IV criteria).
* A group of 30 control subjects with no personal or family history of severe psychiatric disorder (bipolar disorder, schizophrenia or schizoaffective disorder), recruited from the staff of the University Hospital of Reims, the medical faculty of Reims or Marnais center health promotion of Reims, via the intranet and paper display.

The two groups will be matched for age (± 3 years), sex and educational level (± 2 years).

Plan of investigation: the study will be done in two visits:

* The first visit by a psychiatrist for:

  * information on the objectives and the methods of research, verification criteria for inclusion and non-inclusion and participation of obtaining consent (written consent)
  * comprehensive psychiatric evaluation and procurement different scales (anxiety scale, Hamilton depression scale, evaluation of verbal IQ, ...).
* 2nd visit, a maximum of 15 days after the first visit by a psychologist, neuropsychologist for the award of the memories of love and future projections defining self: the experimenter asks the subjects to relate memories 3 and 3 future projections. It is important personal events that arouse strong emotions and that the subjects often think.

Memories and projections reported by the subjects are then classified according to their emotional valence, their content, significance and degree of integration itself.

ELIGIBILITY:
Inclusion Criteria:

BD patients :

* Men or women, right-handed, with a diagnosis of type 1 bipolar disorder, according to the DSM-IV criteria, aged from 18 to 60 years-old
* Native French speaker
* Affiliated to the social security
* Accepting the study after reading the information note and signing the consentment form

Healthy Controls (HC):

* Men or women, right-handed, aged from 18 to 65 years-old
* Native French speaker
* Affiliated to the social security
* Accepting the study after reading the information note and signing the consentment form

Exclusion criteria

BD patients :

* A recent alcohol and/or drug abuse or dependence
* A significant general medical illness, including neurological disorders or head trauma
* A sensorial impairment (visual and/or hearing)

HC:

* A personal or first-degree-relative history of bipolar disorder, schizophrenia or schizoaffective disorder according to DSM-IV
* A recent alcohol and/or drug abuse or dependence
* A significant general medical illness, including neurological disorders or head trauma
* A sensorial impairment (visual and/or hearing)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-05; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
psychological test : Mini International Neuropsychiatric Interview (M.I.N.I.) | Day 01
psychological test : State - Trait Anxiety Inventory Form Y | day 15
psychological test : Hamilton Depression Scale (HAM-D) | Day 01
psychological test : Mill Hill Vocabulary Scale | day 15

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France, France